CLINICAL TRIAL: NCT02118974
Title: Randomized Clinical Trial Comparing Conventional Laparoscopic and Robot-Assisted Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Timothy A Deimling, Fellow Minimally Invasive GYN Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000164
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Menorrhagia; Pelvic Pain; Hysterectomy
Keywords: Hysterectomy; Robot-assisted; Laparoscopy
MeSH Terms: conditions — Menorrhagia; Pelvic Pain | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-assisted (Experimental): Robot-assisted hysterectomy
  Interventions: Procedure: Hysterectomy
- Laparoscopic Hysterectomy (Experimental): Laparoscopic Hysterectomy
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Hysterectomy

SUMMARY:
Robotic-assisted surgery is becoming more prominent within the specialty of Gynecologic surgery with little direct evidence that it is if not better than traditional laparoscopic surgery, at least equivalent. We designed a randomized-controlled trial to compare operative times, length of hospital stay, estimated blood loss, and post-operative complications associated with these two methods of minimally invasive hysterectomy.

DETAILED DESCRIPTION:
The proposed study will be a non-blinded randomized control trial. Patients will be randomized into each group Conventional Laparoscopic Hysterectomy (Group #1) and Robot-Assisted Laparoscopic Hysterectomy (Group #2) using a random number generator. Data collection will occur during the following points of patient interaction: pre-operative appointment, the surgical procedure, the patient's hospitalization, first post-operative appointment, and final post-operative appointment.

The care for the patients enrolled in this study will not deviate from the standard care of patients who are currently undergoing laparoscopic and robot-assisted laparoscopic hysterectomy. The patients who present to the office for pre-operative history and physical examination for laparoscopic hysterectomy will be counseled about participation in this study. Basic data collection will commence at the pre-operative visiting, including: patient demographics, past medical history, past surgical history, physical exam findings, and imaging results. The pre-operative appointment will occur between one to thirty days prior to surgery. Intra-operative and immediate post-operative data will be collected by the surgical assistant (resident or fellow) and will include surgical procedure (conventional laparoscopic or robot-assisted), operative time, hematocrit, estimated blood loss, length of stay, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Hysterectomy
* Able to consent to the procedure

Exclusion Criteria:

1. Medical conditions not allowing for pneumoperitoneum
2. Medical conditions not allowing proper ventilation during anesthesia
3. Pelvic organ prolapse amendable to a vaginal approach
4. Pregnant women
5. Patients undergoing planned combined procedures including bowel resection (other than coincidental appendectomy) or major urologic procedures.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Operative Time | Intra operative
  The primary end point is difference in operative time

SECONDARY OUTCOMES:
Complications | up to 6 weeks following intervention
  Complications related to the procedure including delays in discharge and re-admissions will be monitored and evaluated individually throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deimling TA, Eldridge JL, Riley KA, Kunselman AR, Harkins GJ. Randomized controlled trial comparing operative times between standard and robot-assisted laparoscopic hysterectomy. Int J Gynaecol Obstet. 2017 Jan;136(1):64-69. doi: 10.1002/ijgo.12001. Epub 2016 Nov 3. PMID 28099699